CLINICAL TRIAL: NCT04888000
Title: An Exploratory Study Examining Use of the Oxygen for Caregivers® Program
Brief Title: Interprofessional Group Intervention to Enhance Compassion Satisfaction and Resilience
Acronym: CSRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Colleen J Klein, Education & Research Scientist, OSF Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1684111
Record Dates: First submitted 2021-05-05; First posted 2021-05-17 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Compassion Fatigue; Resilience
Keywords: Compassion Fatigue; Resilience
MeSH Terms: conditions — Compassion Fatigue | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single (Other): Educational intervention.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Professional development program provided to small groups of health care professionals in three different sessions over a period of one month with additional independent individual work to be completed between sessions.

SUMMARY:
The purpose of this study is to evaluate an educational professional development program designed to assist health care professionals in developing self-awareness and self-care choices as a means to avoid compassion fatigue and improve resilience.

DETAILED DESCRIPTION:
Professional caregivers are at risk of compassion fatigue due to the nature of their work and repeated exposure over time to work-related stressors. Symptoms of compassion fatigue may include decreased concentration/productivity, increased sick days, and high turnover rates which directly effect patient satisfaction and safety. Lack of data that supports this use of program, though anecdotally, it has been endorsed and benefits from its use are described. Quality of patient care, workforce engagement, and financial effects from turnover of staff are viewed as negative impacts from compassion fatigue.

Our study seeks to extend the body of knowledge with regard to use of a particular resilience program that has shown some promise in a small pilot study.

ELIGIBILITY:
Inclusion Criteria:

* employment within inpatient or outpatient setting in non-profit healthcare system as a healthcare professional
* Professional direct caregivers (nurses, physicians, advanced practice providers, social workers, counselors, chaplains, respiratory therapists, pharmacists

Exclusion Criteria:

* actively participating in or plans to participate in any other formalized mindfulness-based stress reduction program during the time period of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Professional Quality of Life Scale (ProQOL) Version 5 | Change from baseline compassion fatigue subscale measure at 1 and 6 months assessed by compassion fatigue subscale of ProQOL 5 [ Time Frame: Data collected before the program starts and one month after the end of the program and six months
  Professional Quality of Life Scale (ProQOL) Version 5 Compassion Fatigue Subscale
Professional Quality of Life Scale (ProQOL) Version 5 | Change from baseline burnout subscale measure at 1 and 6 months assessed by burnout subscale of ProQOL 5 [ Time Frame: Data collected before the program starts and one month after the end of the program and six months
  Professional Quality of Life Scale (ProQOL) Version 5 Burnout Subscale
Professional Quality of Life Scale (ProQOL) Version 5 | Change from baseline compassion satisfaction subscale measure at 1 and 6 months assessed by compassion satisfaction subscale of ProQOL 5 [ Time Frame: Data collected before the program starts and one month after the end of the program and six months
  Professional Quality of Life Scale (ProQOL) Version 5 Compassion Satisfaction Subscale
Brief Resilience Scale | Change from baseline in resilience measure at 1 month and 6 months assessed by BRS scale [ Time Frame: Data collected before the program starts and one month after the end of the program and six months
  Resilience will be measured using the Brief Resilience Scale (BRS) a 6-item scale developed by Smith et al.(2008).

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Klein, PhD, MS, RN, Principal Investigator — OSF Healthcare System
Locations (1):
- OSF HealthCare System, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ang SY, Hemsworth D, Uthaman T, Ayre TC, Mordiffi SZ, Ang E, Lopez V. Understanding the influence of resilience on psychological outcomes - Comparing results from acute care nurses in Canada and Singapore. Appl Nurs Res. 2018 Oct;43:105-113. doi: 10.1016/j.apnr.2018.07.007. Epub 2018 Jul 26. PMID 30220356
- [Background] Austin CL, Saylor R, Finley PJ. Moral distress in physicians and nurses: Impact on professional quality of life and turnover. Psychol Trauma. 2017 Jul;9(4):399-406. doi: 10.1037/tra0000201. Epub 2016 Oct 31. PMID 27797570
- [Background] Cavanagh N, Cockett G, Heinrich C, Doig L, Fiest K, Guichon JR, Page S, Mitchell I, Doig CJ. Compassion fatigue in healthcare providers: A systematic review and meta-analysis. Nurs Ethics. 2020 May;27(3):639-665. doi: 10.1177/0969733019889400. Epub 2019 Dec 12. PMID 31829113
- [Background] Fortney L, Luchterhand C, Zakletskaia L, Zgierska A, Rakel D. Abbreviated mindfulness intervention for job satisfaction, quality of life, and compassion in primary care clinicians: a pilot study. Ann Fam Med. 2013 Sep-Oct;11(5):412-20. doi: 10.1370/afm.1511. PMID 24019272
- [Background] Huey CWT, Palaganas JC. What are the factors affecting resilience in health professionals? A synthesis of systematic reviews. Med Teach. 2020 May;42(5):550-560. doi: 10.1080/0142159X.2020.1714020. Epub 2020 Jan 25. PMID 31984844
- [Background] Kelly L, Runge J, Spencer C. Predictors of Compassion Fatigue and Compassion Satisfaction in Acute Care Nurses. J Nurs Scholarsh. 2015 Nov;47(6):522-8. doi: 10.1111/jnu.12162. Epub 2015 Aug 19. PMID 26287741
- [Background] Klein CJ, Riggenbach-Hays JJ, Sollenberger LM, Harney DM, McGarvey JS. Quality of Life and Compassion Satisfaction in Clinicians: A Pilot Intervention Study for Reducing Compassion Fatigue. Am J Hosp Palliat Care. 2018 Jun;35(6):882-888. doi: 10.1177/1049909117740848. Epub 2017 Nov 23. PMID 29169248
- [Background] McKinley N, Karayiannis PN, Convie L, Clarke M, Kirk SJ, Campbell WJ. Resilience in medical doctors: a systematic review. Postgrad Med J. 2019 Mar;95(1121):140-147. doi: 10.1136/postgradmedj-2018-136135. Epub 2019 Mar 29. PMID 30926716
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Potter P, Deshields T, Berger JA, Clarke M, Olsen S, Chen L. Evaluation of a compassion fatigue resiliency program for oncology nurses. Oncol Nurs Forum. 2013 Mar;40(2):180-7. doi: 10.1188/13.ONF.180-187. PMID 23448743